CLINICAL TRIAL: NCT05856617
Title: Comparison of Remimazolam and Propofol as an Induction Agent for Morbid Obesity Patients Undergoing Laparoscopic Sleeve Gastrectomy
Brief Title: Remimazolam vs Propofol as an Induction Agent for Morbid Obesity Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, In-Ae Song, Associate professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B-2208-774-001
Record Dates: First submitted 2023-05-03; First posted 2023-05-12 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Remimazolam; Desflurane; Morbid Obesity; Sleeve Gastrectomy; General Anesthesia
Keywords: Remimazolam; Desflurane; Morbid obesity; sleeve gastrectomy
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Who Masked: Participant
Masking Description: Did not tell them about assigned group till all the measurement ends.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remimazolam (Experimental): Anesthesia induction with remimazolam
  Interventions: Drug: Remimazolam besylate
- Propofol (No Intervention): Anesthesia induction with propofol

INTERVENTIONS:
Drug: Remimazolam besylate — Remimazolam besylate anesthesia induction
  Arms: Remimazolam

SUMMARY:
It is known that morbidly obese patients are often accompanied by cardiovascular complications such as hypertension, cardiac hypertrophy, and diastolic dysfunction, and are known to increase the risk of hypotension during anesthesia induction. Remimazolam is widely used in Japan and the United States, and it was approved as a drug for general anesthesia and sedation in Korea in 2021. It was reported that remimazolam caused less hypotension after induction of anesthesia than propofol. However, there is no study on the use of remimazolam in patients undergoing bariatric surgery due to morbid obesity. Therefore, through this study, we plan to check whether remimazolam is safe and effective as an anesthetic-inducing agent for morbidly obese patients undergoing bariatric surgery.

DETAILED DESCRIPTION:
According to a report by M.Doi et al., the incidence of hypotension was 20% in the group using remimazolam 6mg/kg/hr as an anesthetic induction dose for surgical patients, which was significantly higher than that of the control group using propofol (49.3%). When the number of subjects was calculated by a two-sided significance test with an alpha error rate of 0.05 and a power of 80% (experimental group 20%, control group 49.3%; chi square), each group required 40 subjects considering the following. With dropout rate of 10%, total of 44 subjects in each group were required.

Among the patients who were admitted to Seoul National University Bundang Hospital and underwent laparoscopic sleeve gastrectomy under general anesthesia, patients who voluntarily signed the consent form after listening to sufficient explanations about this clinical trial and taking sufficient time to make a decision were eligible. The explanation of consent is provided by the medical staff (doctor), such as the principal researcher or co-researcher of this study, and when the consent form is signed, the person is listed as a research subject. There is no separate pre-screening other than taking a medical history for research subject selection.

We will do the modified intention-to-treat group analysis, which means that we will include all cases except for cases that the subject was found major selection criteria were violated after assignment of subject numbers, cases that administration of investigational drugs was not initiated, or cases where major data about efficacy can not be obtained after medication administration initiation in analyses. Additionally we will report excluded cases with the exclusion reasons.

Statistical analysis

* Tested by analyzing the t-test of the mean value test (the Mann-Whitney U test when normality is not satisfied) when normality is satisfied in the case of non-scale according to the scale of the outcome variable In the case of a chi-squared categorical variable (expected frequency is 20 % less than 5 cells and analyzed using Fisher's exact test), or Fisher's exact test (when it is possible).
* If the P value is less than 0.05, it is judged as a significant result.

Handling missing data

- Missing values from this test will not be replaced unless otherwise specified.

ELIGIBILITY:
Inclusion Criteria:

* =or > 20 years
* Admission for General anesthesia for sleeve gastrectomy

Exclusion Criteria:

* No severe adverse effect history or hypersensitivity of benzodiazepines or its additives
* Acute alcoholic intoxication state
* Coma or shock state due to other condition than heart problem.
* Acute narrow-angle glaucoma

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2022-10-25 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-09-12 (Estimated)

PRIMARY OUTCOMES:
Rate of hypotension event | During anesthesia induction
  Hypotension event

SECONDARY OUTCOMES:
Induction time | During anesthesia induction
  Induction dose administration~LOC
Vasopressor (total amount) | During anesthesia induction
  Total ephedrine dose

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul national university Bundang hospital, Seongnam-si, South Korea